CLINICAL TRIAL: NCT07114198
Title: Pain Management in Teeth With Reversible Pulpitis: A Randomised Controlled Trial
Brief Title: Pain Management in Teeth With Reversible Pulpitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Merve Bilmez Selen, Dr. lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethics number:2024-KAEK-08
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Reversible Pulpitis; Ibuprofen
Keywords: reversible pulpitis; ibuprofen; dental pain
MeSH Terms: conditions — Toothache | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Children in this group received no preoperative medication before undergoing vital pulp therapy. Standard local anesthesia was administered prior to the procedure.
- ibuprofen group (Experimental): Children in this group received a single dose of ibuprofen (10 mg/kg) orally, 40 minutes prior to vital pulp therapy. The goal was to evaluate the effect of preoperative ibuprofen on intraoperative pain and physiological stress.
  Interventions: Drug: Ibuprofen 10 mg/kg

INTERVENTIONS:
Drug: Ibuprofen 10 mg/kg — Ibuprofen was administered orally at a dose of 10 mg/kg body weight, 40 minutes before the start of the dental procedure. This intervention was designed to reduce intraoperative pain and pulse elevation associated with reversible pulpitis.
  Arms: ibuprofen group

SUMMARY:
Effective intraoperative pain management is vital in paediatric dentistry, especially during vital pulp therapy (VPT) for reversible pulpitis. Although NSAIDs are widely used postoperatively, their role in controlling pain during treatment is less understood. To investigate the effect of preoperative ibuprofen on pain perception and physiological stress during VPT in children.

DETAILED DESCRIPTION:
This prospective, randomized, controlled clinical trial will investigate the effect of preoperative ibuprofen administration on intraoperative pain during vital pulp therapy (VPT) in pediatric patients diagnosed with reversible pulpitis. The study will be conducted at the Department of Pediatric Dentistry, Faculty of Dentistry, Inonu University. Ethical approval has been obtained from the Institutional Clinical Research Ethics Committee of Inonu University (Approval No: 2024-KAEK-08; Date: 25.12.2024). Written informed consent will be obtained from the parents of all participants.

A total of 44 children aged 7 to 13 years, in good general health, with deep carious lesions in a mandibular first permanent molar and a clinical diagnosis of reversible pulpitis will be included in the study. Participants will be randomly assigned in equal numbers (n=22 per group) to the intervention and control groups using a computer-generated randomization sequence and the sealed envelope method.

Children in the intervention group will receive oral ibuprofen (10 mg/kg) 40 minutes prior to treatment. The control group will receive no preoperative medication. A single-blind study design will be employed: the clinician performing the procedures will be aware of group allocation, while the statistician responsible for data analysis will remain blinded.

All participants will receive an inferior alveolar nerve block (IANB) before the procedure. Anesthesia will be verified with a cold test, and treatment will begin only after adequate anesthesia is confirmed. All procedures will be performed by the same pediatric dentist, following a standardized clinical protocol. The specific type of VPT (protective liner, direct pulp capping, partial pulpotomy, or coronal pulpotomy) will be selected based on clinical presentation.

Intraoperative pain will be assessed using both physiological and subjective measures. Pulse rate will be continuously monitored with a fingertip pulse oximeter, with a focus on readings taken when the bur approaches within close proximity to the pulp. Subjective pain will be measured using a Visual Analogue Scale (VAS), shown to the patient at the most sensitive moment of the procedure. Postoperative VAS scores will be recorded on Days 1, 3, and 7.

ELIGIBILITY:
Inclusion Criteria:

* Children with no history of systemic disease,
* Demonstrated cooperative behaviour during treatment,
* Parental consent obtained for study participation,
* Presence of a first permanent mandibular molar with:

  1. Clinical and radiographic diagnosis of reversible pulpitis,
  2. Deep carious lesion extending beyond three-quarters of dentine thickness on periapical/bitewing radiographs (ICDAS score 5-6),
  3. Positive cold test response with Endo-Ice (Hygienic Corp., Akron, OH, USA) producing short-lasting pain (subsiding within <10 seconds after stimulus removal),
  4. No clinical signs of swelling, abscess, or sinus tract,
  5. Absence of abnormal tooth mobility,
  6. Restorability of the tooth.

Exclusion Criteria:

* Presence of primary teeth requiring treatment,
* Clinical or radiographic diagnosis of irreversible pulpitis, necrotic pulp, apical lesion, swelling, abscess, or sinus tract,
* Analgesic intake within the preceding 12 hours,
* Known allergy to ibuprofen or local anaesthetics,
* Neurological or psychiatric developmental disorders,
* Presence of systemic illness,
* Existing gastrointestinal disease.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2025-08-02 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want it because the work hasn't been completed yet.

REFERENCES:
- [Result] Carrasco-Labra A, Polk DE, Urquhart O, Aghaloo T, Claytor JW Jr, Dhar V, Dionne RA, Espinoza L, Gordon SM, Hersh EV, Law AS, Li BS, Schwartz PJ, Suda KJ, Turturro MA, Wright ML, Dawson T, Miroshnychenko A, Pahlke S, Pilcher L, Shirey M, Tampi M, Moore PA. Evidence-based clinical practice guideline for the pharmacologic management of acute dental pain in children: A report from the American Dental Association Science and Research Institute, the University of Pittsburgh School of Dental Medicine, and the Center for Integrative Global Oral Health at the University of Pennsylvania. J Am Dent Assoc. 2023 Sep;154(9):814-825.e2. doi: 10.1016/j.adaj.2023.06.014. PMID 37634915
- [Result] Shirvani A, Shamszadeh S, Eghbal MJ, Marvasti LA, Asgary S. Effect of preoperative oral analgesics on pulpal anesthesia in patients with irreversible pulpitis-a systematic review and meta-analysis. Clin Oral Investig. 2017 Jan;21(1):43-52. doi: 10.1007/s00784-016-1974-1. Epub 2016 Nov 11. PMID 27837343
- [Result] Pozzi A, Gallelli L. Pain management for dentists: the role of ibuprofen. Ann Stomatol (Roma). 2011 Jul;2(3-4 Suppl):3-24. Epub 2012 Apr 15. No abstract available. PMID 22888399
- [Result] Hargreaves K, Abbott PV. Drugs for pain management in dentistry. Aust Dent J. 2005 Dec;50(4 Suppl 2):S14-22. doi: 10.1111/j.1834-7819.2005.tb00378.x. PMID 16416713
- See also: ADA-Evidence-based clinical practice guideline for the pharmacologic management of acute dental pain in children. — https://doi.org/10.1016/j.adaj.2023.06.014
- See also: Related Info — https://doi.org/10.1016/j.adaj.2023.06.014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 children were enrolled in the study. Participants were randomized into two groups (23 in the control group, 23 in the ibuprofen group). Two participants did not complete the study due to protocol violations, leaving 44 participants who completed the trial.
Pre-assignment Details: Randomization was performed using a sealed envelope method; the envelope contents were prepared by a third researcher before the examination. Because double-blinding was not possible, a single-blind design was employed. The clinician performing the procedure was aware of the groups, but the statistician performing the data analysis was unaware of the groups.
Period: Overall Study
Arm/Group | Control Group | Ibuprofen Group
Started | 23 (23 PATIENTS WERE INCLUDED IN THIS GROUP) | 23 (23 PATIENTS WERE INCLUDED IN THIS GROUP)
Completed | 22 (22 PATIENTS WERE INCLUDED IN THIS GROUP.) | 22 (22 PATIENTS WERE INCLUDED IN THIS GROUP.)
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who met the inclusion criteria and had baseline demographic data available were included in this analysis. One participant from each group was excluded due to protocol violation, leaving 22 participants per group (total n=44).
Groups:
- Control Group: Children in this group received no preoperative medication before undergoing vital pulp therapy. Standard local anesthesia was administered prior to the procedure.The mean age of participants was 9.32 years (SD ±1.96). The group consisted of 16 females (72.7%) and 6 males (27.3%).
- Ibuprofen Group: Children in this group received a single dose of ibuprofen (10 mg/kg) orally, 40 minutes prior to vital pulp therapy. The goal was to evaluate the effect of preoperative ibuprofen on intraoperative pain and physiological stress.
  Ibuprofen 10 mg/kg: Ibuprofen was administered orally at a dose of 10 mg/kg body weight, 40 minutes before the start of the dental procedure. This intervention was designed to reduce intraoperative pain and pulse elevation associated with reversible pulpitis.The mean age of participants was 9.59 years (SD ±1.56). The group consisted of 14 females (63.6%) and 8 males (36.4%).
- Total: Total of all reporting groups
Arm/Group | Control Group | Ibuprofen Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 22 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was measured in years at the time of enrollment and is reported as a continuous variable (mean ± standard deviation).
  years | 9.32 (1.96) | 9.59 (1.76) | 9.45 (1.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 6 | 8 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — All participants were of the same ethnic background (Turkish).
  Participants
    Turkish | 22 | 22 | 44
Region of Enrollment [Number; unit: participants] — All participants were recruited from Turkey. Population: TURKEY
  participants
    Turkey | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity From Baseline (Pre-Operative) to Immediately During the Procedure (Day 0), Measured by the Visual Analogue Scale (VAS)
Description: Pain intensity will be assessed using the Visual Analogue Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). The change will be calculated as the score immediately during the procedure (Day 0) minus the Baseline (Pre-Operative) score. Higher scores indicate worse pain.
Time Frame: Pre-Operative (Baseline) and Immediately During the Procedure (Day 0)
Population: 7-13 years children
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Ibuprofen Group
Number analyzed (Participants) | 22 | 22
score on a scale | 5.05 (3.51) | 0.64 (1.14)

2. Secondary Outcome: Change in Postoperative Pain Intensity From Baseline (Pre-Operative) to Day 1, Measured by the Visual Analogue Scale (VAS)
Description: Pain intensity will be assessed using the Visual Analogue Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). The Baseline (Pre-Operative) VAS score will be compared with the VAS score reported by the participant on Day 1. On Day 1, participants will be contacted by phone and asked to rate their pain using the same VAS tool.
Time Frame: Pre-Operative (Baseline) and 1 days post-treatment (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Ibuprofen Group
Number analyzed (Participants) | 22 | 22
score on a scale | 0.59 (1.37) | 0.68 (1.39)

3. Other Pre Specified Outcome: Change in Postoperative Pain Intensity From Baseline (Pre-Operative) to Day 7, Measured by the Visual Analogue Scale (VAS)
Description: Pain intensity will be assessed using the Visual Analogue Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). The Baseline (Pre-Operative) VAS score will be compared with the VAS score reported by the participant on Day 3. On Day 3, participants will be contacted by phone and asked to rate their pain using the same VAS tool.
Time Frame: Pre-Operative (Baseline) and 3 days post-treatment (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Ibuprofen Group
Number analyzed (Participants) | 22 | 22
score on a scale | 0.14 (0.47) | 0.23 (0.75)

4. Other Pre Specified Outcome: Change in Postoperative Pain Intensity From Baseline (Pre-Operative) to Day 7, Measured by the Visual Analogue Scale (VAS)Analogue Scale (VAS)
Description: Pain intensity will be assessed using the Visual Analogue Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). The Baseline (Pre-Operative) VAS score will be compared with the VAS score reported by the participant on Day 7. On Day 7, participants will be contacted by phone and asked to rate their pain using the same VAS tool.
Time Frame: Pre-Operative (Baseline) and 7 days post-treatment (Day 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Ibuprofen Group
Number analyzed (Participants) | 22 | 22
score on a scale | 0.05 (0.21) | 0.09 (0.29)

ADVERSE EVENTS:
Time Frame: two weeks
Description: Adverse events were monitored in all participants at risk (n=22 per group; total 44). No all-cause mortality events were observed. All-Cause Mortality, Serious Adverse Events, and Other (Non-Serious) Adverse Events were not monitored or assessed in this study; therefore, the number of participants at risk is 0.
Groups:
- Control Group: Children in this group received no preoperative medication before undergoing vital pulp therapy. Standard local anesthesia was administered prior to the procedure.
  Patients who did not receive ibuprofen after the procedure (N=22
- Ibuprofen Group: Children in this group received a single dose of ibuprofen (10 mg/kg) orally, 40 minutes prior to vital pulp therapy. The goal was to evaluate the effect of preoperative ibuprofen on intraoperative pain and physiological stress.
  Ibuprofen 10 mg/kg: Ibuprofen was administered orally at a dose of 10 mg/kg body weight, 40 minutes before the start of the dental procedure. This intervention was designed to reduce intraoperative pain and pulse elevation associated with reversible pulpitis.Patients who received ibuprofen after the procedure (N=22).
Arm/Group | Control Group | Ibuprofen Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT07114198/Prot_SAP_000.pdf